CLINICAL TRIAL: NCT02369614
Title: Low-Frequency Versus High-Frequency Repetitive Transcranial Magnetic Stimulation of the Right Dorsolateral Prefrontal Cortex in Posttraumatic Stress Disorder
Brief Title: Low -vs- High-Frequency Repetitive TMS of the Right Dorsolateral Prefrontal Cortex in PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing issues
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Donald Hurst, LCDR Donald Hurst, MD, MC USN, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NMCSD.2014.0061
Record Dates: First submitted 2014-11-17; First posted 2015-02-24 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: rTMS - repetitive transcranial magnetic stimulation; CAPS - Clinician Administered PTSD Scale
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active Comparator:1 Hz rTMS (Active Comparator): Active Comparator: 1 Hz rTMS
  Interventions: Other: Active Comparator: 1 Hz rTMS
- Active Comparator:10 Hz rTMS (Active Comparator): Active Comparator:10 Hz rTMS
  Interventions: Other: Active Comparator: 10 Hz rTMS
- Sham Comparator:Sham rTMS (Sham Comparator): Sham Comparator: Sham rTMS
  Interventions: Other: Sham Comparator:
- OASIS treatment as usual (No Intervention): OASIS treatment as usual

INTERVENTIONS:
Other: Active Comparator: 1 Hz rTMS — 1 Hz rTMS
  Arms: Active Comparator:1 Hz rTMS
Other: Active Comparator: 10 Hz rTMS — 10 Hz rTMS
  Arms: Active Comparator:10 Hz rTMS
Other: Sham Comparator: — Sham rTMS
  Arms: Sham Comparator:Sham rTMS

SUMMARY:
This is a randomized placebo/sham controlled, double-blind study investigating the efficacy of high- and low-frequency rTMS applied to the right DLPFC at either 1 Hz, 10 Hz, or sham rTMS as compared to an OASIS treatment as usual group for the treatment of PTSD symptoms.

DETAILED DESCRIPTION:
The study will be carried out within the Overcoming Adversity and Stress Injury Support (OASIS) program administered by Naval Medical Center San Diego (NMSD). OASIS is a residential treatment program developed for active duty service members diagnosed with combat related PTSD. OASIS is a 9 week program in which cohorts of 10 patients undergo a variety of therapeutic activities with a focus on cognitive processing therapy (CPT) of combat trauma conducted in both group and individual formats.

Subjects who qualify will be assigned by block randomization to one of four arms:

1. 1 Hz rTMS of the right dorsolateral prefrontal cortex
2. 10 Hz rTMS of the right dorsolateral prefrontal cortex
3. Sham rTMS of the right dorsolateral prefrontal cortex
4. OASIS treatment as usual

Treatment will be administered in 10 daily sessions, conducted on weekdays, for 2 consecutive weeks. .

ELIGIBILITY:
Inclusion Criteria:

Participant in the OASIS program

Willing and able to give informed consent

Diagnosis of Post-Traumatic Stress Disorder as determined by the CAPS CAPS score of at least 50

Males or females between 18-65 years of age

Exclusion Criteria:

Current primary Axis I disorder including Schizophrenia, Bipolar Disorder type I, Active Substance use

Patients with severe or unstable medical conditions, which in the opinion of the investigator would interfere with their progress or safety

ECT treatment within the last 30 days Patients with neurological disorder leading to increased intracranial pressure

Participation in other interventional treatment protocols (participants of monitoring/observational studies can be included)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in Clinician Administered PSTD Scale (CAPS) score from Baseline to week 4 | Baseline and Week 4
  Clinician Administered PSTD Scale (CAPS)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Hurst, MD, Principal Investigator — NMCSD

IPD SHARING:
Plan to Share IPD: No